CLINICAL TRIAL: NCT02282579
Title: Spanish Retrospective Study to Evaluate the Efficacy and Safety of Targeted Therapies After Pazopanib as First-line Therapy, in Patients With Metastatic Renal Cell Carcinoma in Daily Clinical Practice
Brief Title: Spanish Retrospective Study to Evaluate the Efficacy and Safety of Targeted Therapies After Pazopanib as First-line Therapy
Acronym: SPAZO
Status: Completed | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Other Study IDs: SOG-SPA-2014-02
Record Dates: First submitted 2014-09-10; First posted 2014-11-04 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient with metastatic renal cell carcinoma treated: Patient with metastatic renal cell carcinoma treated with Pazopanib
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Non interventional study

SUMMARY:
The purpose of this retrospective observational study was to analyze the effect of targeted therapies administered as second-line treatment after failure of pazopanib as well as increase the amount of information available on efficacy and safety of pazopanib as a first-line therapy in practice usual for the clinical treatment of metastatic Renal Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18.
* Metastatic renal cell cancer of any histology.
* Patients treated with pazopanib for metastatic cell renal cancer outside the context of clinical trials (clinical practice) in Spanish centers from 1 April 2011 until 30 June 2014. shall be included all patients who received pazopanib as first-line treatment in each participating center, whether had experienced treatment failure with pazopanib or were still in first-line treatment. The inclusion of patients who are also allowed received cytokine as first-line treatment followed by pazopanib as well as patients who received sunitinib as first-line treatment and have changed pazopanib for toxicity or intolerance, provided they have not received more a cycle of sunitinib.
* Centers that agree to participate must commit to: · Include all patients meeting the inclusion criteria to reduce by possible selection bias. Because it supplies only pazopanib Hospital pharmacy service (not outside hospitals), the identification of patients will be performed at the hospital pharmacy records in each participating center.

Exclusion Criteria:

* Patients who received pazopanib in clinical trials or treatment second line, with the exceptions noted above.
* Patients with the diagnosis and / or treatment of malignancies of importance other than Cell renal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is aimed at patients who received pazopanib in first-line metastatic cell renal cancer, so care (clinical trial patients are excluded) in the period from April 2011 (date of approval of pazopanib in Spain) to 30 June 2014, ie, before the presentation of CEICs in each hospital. In all cases, any decision to administer pazopanib therapy in first line will be taken according to local clinical practice and prior to the inclusion of patients in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Describe the efficacy in terms of response | 3 years
  Describe the efficacy in terms of response of second-line targeted therapies administered in patients with metastatic clear cell carcinoma treated pazopanib as a first-line therapy in routine clinical practice (unselected population).
Describe the efficacy in terms of progression-free survival (PFS) | 3 years
  Describe the efficacy in terms of progression-free survival (PFS) of second-line targeted therapies administered in patients with metastatic clear cell carcinoma treated pazopanib as a first-line therapy in routine clinical practice (unselected population).
Describe the efficacy in terms of overall survival (OS) | 3 years
  Describe the efficacy in terms of overall survival (PFS) of second-line targeted therapies administered in patients with metastatic clear cell carcinoma treated pazopanib as a first-line therapy in routine clinical practice (unselected population).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Arranz, PhD, Principal Investigator — Investigator coordinator
Locations (34):
- Spain (34):
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Vall d' Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital G U de Ciudad Real, Ciudad Real
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital San Cecilio, Granada
  - Hospital General Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital de León, León
  - Hospital San Pedro Logroño, Logroño
  - Hospital Lucus Augusti, Lugo
  - Hospital Gregorio Marañon, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Quirón, Madrid
  - Hospital U Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Provincial de Pontevedra, Pontevedra
  - Hospital Clínico Universitario Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Marques de Valdecilla, Santander
  - Hospital Ntra. Sra. De Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico de Valencia, Valencia
  - Hospital Gral Universitario Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - IVO Valencia, Valencia
  - Hospital Rio Hortega, Valladolid
  - CHUVI ( Vigo), Vigo
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza